CLINICAL TRIAL: NCT00465075
Title: An Open-Label, Single-Dose, 3-Period, Crossover Study To Determine The Effect Of A High-Fat Meal On The Relative Bioavailability And Pharmacokinetics Of A Single Dose Of Bazedoxifene Acetate/Conjugated Estrogens (Premarin© New Process) Administered Orally To Healthy, Postmenopausal Women
Brief Title: Study Evaluating Bazedoxifene/Conjugated Estrogens Combinations in Fed and Fasting in Healthy, Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 3115A1-1116
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Healthy
MeSH Terms: interventions — bazedoxifene

INTERVENTIONS:
Drug: Bazedoxifene/conjugated estrogens combination

SUMMARY:
The primary objective is to determine the effect of a high-fat meal on the bioavailability and PK of a single, oral dose of BZA/CE (PNP) 20mg/0.625 strength tablet, assessing both the BZA and CE components.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by the investigator on the basis of history, physical examinations, clinical laboratory test results, vital signs, and 12-lead ECGs.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2007-03; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
PK parameters

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Gainesville, Florida, United States